CLINICAL TRIAL: NCT07086547
Title: The Effect of Education Provided With Artificial Intelligence-Based Materials on Mothers' Fever Management and Anxiety Levels
Brief Title: Impact of Artificial Intelligence-Supported Educational Intervention on Mothers' Fever Management
Acronym: AI-FEVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISMIRA JULFAYEVA (Other)
Responsible Party: Sponsor-Investigator, ISMIRA JULFAYEVA, Master's Student and nurse, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10718356; 10718356 (Other: Erciyes University, Institute of Health Sciences)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fever; Pediatric Fever Management; Parental Anxiety
Keywords: Fever, Pediatric Fever, Fever Management, Parental Education, Anxiety, Artificial Intelligence, AI Education, Child Health, Clinical Trial
MeSH Terms: conditions — Fever; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants (mothers of children) will be randomly assigned to one of two groups: an intervention group receiving AI-supported fever management education, and a control group receiving standard care. Outcomes will be compared between the two groups to evaluate the effect of the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Based Education Group (Experimental): Mothers in this group will receive fever management education developed using an artificial intelligence language model (ChatGPT 4.0). The education includes written materials with visual content on managing fever in children and is delivered as a one-time structured session.
  Interventions: Other: AI-Based Fever Management Education
- Control Group (No Intervention): Mothers in this group will receive routine care and no additional fever education materials.

INTERVENTIONS:
Other: AI-Based Fever Management Education — This intervention consists of a fever management education program developed using ChatGPT 4.0, a large language model by OpenAI. The educational content includes seven pages and eight visuals explaining how to manage fever in children. The content was reviewed by pediatric specialists and revised accordingly. It is delivered as a one-time structured session to mothers in the intervention group.
  Other Names: ChatGPT-based Educational Material
  Arms: AI-Based Education Group

SUMMARY:
This study aims to evaluate the effect of an artificial intelligence (AI)-based educational program on mothers' knowledge and anxiety related to fever management in children. Fever is a common symptom in pediatric patients, especially under the age of three, causing repeated health concerns for parents. Despite the prevalence of fever, parents often lack sufficient knowledge and skills to manage it properly, which may lead to unnecessary anxiety and inappropriate care practices.

The study will be conducted as a pretest-posttest experimental design including 80 mothers of children who visit the Pediatric Emergency Clinic at Kayseri City Hospital. Participants will be assigned to either an intervention group receiving AI-supported fever management education or a control group receiving standard care.

Data will be collected using validated scales to assess parental fever management knowledge and anxiety levels before and after the intervention. The educational material was developed using ChatGPT 4.0, a large language model AI platform, and reviewed by pediatric experts.

The results of this study may improve fever management education and reduce anxiety among mothers, potentially leading to better health outcomes for children.

DETAILED DESCRIPTION:
This study investigates the impact of an AI-supported educational program on mothers' fever management knowledge and anxiety. Fever is common in pediatric patients and can cause significant concern for parents, especially for children under three years old. Parents often lack adequate knowledge about fever management, leading to inappropriate practices and increased anxiety.

The study uses a pretest-posttest experimental design involving 80 mothers visiting the Pediatric Emergency Clinic at Kayseri City Hospital. Participants are assigned to either an intervention group receiving education developed using ChatGPT 4.0, reviewed by pediatric experts, or a control group receiving standard care.

Data collection tools include validated scales measuring fever management knowledge and anxiety levels. The intervention aims to empower mothers with better skills and reduce anxiety, potentially improving child health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged over 18 years,
* Mothers with children aged between 6 months and 5 years,
* No hearing problems,
* Agree to participate in the study,
* Presenting to the pediatric emergency department with a complaint of fever in their child,
* Child admitted to the emergency observation room for treatment,
* Able to speak and understand Turkish.

Exclusion Criteria:

* Illiterate mothers,
* Mothers whose children have had febrile seizures,
* Mothers whose children have comorbid diseases,
* Mothers whose children have symptoms requiring medical intervention other than fever.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Fever Management Practices | Baseline and 2 weeks after intervention
  Measured using the Parental Fever Management Scale. The difference between pre- and post-intervention scores will be analyzed.
Change in Parental Fever Management Practices | Baseline and 2 weeks after intervention
  Measured using the Parental Fever Management Scale. Higher scores indicate better fever management practices. The change from baseline to post-intervention will be assessed.

SECONDARY OUTCOMES:
Change in Parental Anxiety Levels | Baseline and 2 weeks after intervention
  Measured using the short version of the State Anxiety Inventory (STAI). A decrease in the score indicates reduced anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University (ERÜ) Health Application and Research Center, Fevzi Mercan-Mustafa Eraslan Children's Hospital, Pediatric Emergency Unit, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
"We have not yet determined whether individual participant data will be shared. Decisions will be made after study completion."